CLINICAL TRIAL: NCT04108416
Title: Unilateral Cleft Repair in One Surgery With Pure Primary Healing
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Benito Benitez, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: PurePrimary
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cleft Lip and Palate
Keywords: cleft lip; cleft palate; cleft lip and palate; orofacial cleft
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cleft lip and palate repair — The intervention is the currently used cleft lip and palate repair technique at the University Hospital Basel and University Childrens Hospital Basel

SUMMARY:
Retrospective analysis of the current surgical method to repair unilateral cleft lip and palate malformations at our centre

ELIGIBILITY:
Inclusion Criteria:

* newborn patients with complete unilateral cleft lip and palate

Exclusion Criteria:

* with associated syndrome
* previous lip/ palate repair
* previous presurgical orthopaedics other than passive palatal plate

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn patients with complete unilateral cleft lip and palate treated at the University Hospital Basel in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Cleft size measurement | Measured on a model after birth and at surgery with 8 month of age
  Cleft size is measured before and after passive palatal plate therapy

SECONDARY OUTCOMES:
Wound healing | 1, 3 and 6 month after surgery
  Full primary healing of the former cleft, no fistula formation, no oronasal leaking
Adverse events | 6 month
  Surgical and anaesthesia-relate adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Benitez Benito, MD DMD, Principal Investigator — University of Basel and University Hospital Basel
Locations (1):
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
without further approval by our ethical commission individual participant data is not available to other researchers

REFERENCES:
- [Background] Aduss H, Pruzansky S. Width of cleft at level of the tuberosities in complete unilateral cleft lip and palate. Plast Reconstr Surg. 1968 Feb;41(2):113-23. doi: 10.1097/00006534-196802000-00003. No abstract available. PMID 4873510
- [Background] Berkowitz S, Duncan R, Evans C, Friede H, Kuijpers-Jagtman AM, Prahl-Anderson B, Rosenstein S. Timing of cleft palate closure should be based on the ratio of the area of the cleft to that of the palatal segments and not on age alone. Plast Reconstr Surg. 2005 May;115(6):1483-99. doi: 10.1097/01.prs.0000161673.31770.23. PMID 15861051
- [Background] Mueller AA, Zschokke I, Brand S, Hockenjos C, Zeilhofer HF, Schwenzer-Zimmerer K. One-stage cleft repair outcome at age 6- to 18-years -- a comparison to the Eurocleft study data. Br J Oral Maxillofac Surg. 2012 Dec;50(8):762-8. doi: 10.1016/j.bjoms.2012.02.002. Epub 2012 May 1. PMID 22551772
- [Background] Brief J, Behle JH, Stellzig-Eisenhauer A, Hassfeld S. Precision of landmark positioning on digitized models from patients with cleft lip and palate. Cleft Palate Craniofac J. 2006 Mar;43(2):168-73. doi: 10.1597/04-106.1. PMID 16526922
- [Derived] Benitez BK, Brudnicki A, Surowiec Z, Singh RK, Nalabothu P, Schumann D, Mueller AA. Continuous circular closure in unilateral cleft lip and plate repair in one surgery. J Craniomaxillofac Surg. 2022 Jan;50(1):76-85. doi: 10.1016/j.jcms.2021.07.002. Epub 2021 Aug 3. PMID 34896005